CLINICAL TRIAL: NCT00644228
Title: A Randomized Phase III Trial of CC-5013 (Lenalidomide, NSC-703813) and Low Dose Dexamethasone (LLD) Versus Bortezomib (PS-341, NSC-681239), Lenalidomide And Low Dose Dexamethasone (BLLD) for Induction, in Patients With Previously Untreated Multiple Myeloma Without an Intent for Immediate Autologous Stem Cell Transplant
Brief Title: Lenalidomide and Dexamethasone With or Without Bortezomib in Treating Patients With Previously Untreated Multiple Myeloma
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00798; NCI-2009-00798 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); SWOG-S0777; S0777; CDR0000590321; S0777 (Other: SWOG); S0777 (Other: CTEP); U10CA032102 (NIH); U10CA180888 (NIH)
Record Dates: First submitted 2008-03-22; First posted 2008-03-26 (Estimated); Results first posted 2017-07-06 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-10

CONDITIONS: DS Stage I Multiple Myeloma; DS Stage II Multiple Myeloma; DS Stage III Multiple Myeloma
MeSH Terms: interventions — Bortezomib; Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (dexamethasone and lenalidomide) (Active Comparator): Patients receive dexamethasone PO QD on days 1, 8, 15, and 22 and lenalidomide PO QD on days 1-21. Treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Dexamethasone; Other: Laboratory Biomarker Analysis; Drug: Lenalidomide
- Arm II (dexamethasone, lenalidomide, bortezomib) (Experimental): Patients receive dexamethasone PO QD on days 1, 2, 4, 5, 8, 9, 11, and 12; lenalidomide PO QD on days 1-14; and bortezomib IV over 3-5 seconds on days 1, 4, 8, and 11. Treatment repeats every 21 days for 8 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Bortezomib; Drug: Dexamethasone; Other: Laboratory Biomarker Analysis; Drug: Lenalidomide

INTERVENTIONS:
Drug: Bortezomib — Given IV
  Other Names: [(1R)-3-Methyl-1-[[(2S)-1-oxo-3-phenyl-2-[(pyrazinylcarbonyl)amino]propyl]amino]butyl]boronic Acid; LDP 341; LDP-341; LDP341; MLN 341; MLN-341; MLN341; PS 341; PS-341; PS341; Velcade
  Arms: Arm II (dexamethasone, lenalidomide, bortezomib)
Drug: Dexamethasone — Given PO
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycadron; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decadron DP; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasone Intensol; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Dxevo; Fluorodelta; Fortecortin; Gammacorten; Hemady; Hexadecadrol; Hexadrol; LenaDex; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; TaperDex; Visumetazone; ZoDex
Other: Laboratory Biomarker Analysis — Optional correlative studies
Drug: Lenalidomide — Given PO
  Other Names: CC 5013; CC-5013; CC5013; CDC 501; Revlimid

SUMMARY:
This randomized phase III trial studies lenalidomide, dexamethasone, and bortezomib to see how well it works compared to dexamethasone and lenalidomide alone in treating patients with previously untreated multiple myeloma. Biological therapies, such as lenalidomide, may stimulate the immune system in different ways and stop cancer cells from growing. Drugs used in chemotherapy, such as dexamethasone, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Bortezomib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth or by blocking blood flow to the cancer. It is not yet known whether lenalidomide and dexamethasone is more effective with or without bortezomib in treating multiple myeloma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare progression-free survival (PFS) in patients with newly diagnosed myeloma treated with lenalidomide plus low dose dexamethasone versus bortezomib plus lenalidomide and low dose dexamethasone.

SECONDARY OBJECTIVES:

I. Assess response using the new international response criteria. II. To bank specimens for future translational medicine research. III. Follow patients to assess overall survival and other long-term outcomes stratified by intent to transplant at progression.

TERTIARY OBJECTIVES:

I. To evaluate custom and genome-wide single nucleotide polymorphisms in correlation with biology, prognosis and outcome for both treatment regimens combined; to verify the findings recently obtained with the custom Bank on a Cure program (BOAC) single nucleotide polymorphism (SNP) chip on Total Therapy 2 (TT2) data with respect to bone disease in the cooperative group setting.

II. To use baseline gene expression profiling as a tool to evaluate the biology, prognostic and risk factors, and response to therapy for both treatment regimens combined. To validate John Shaughnessy's 70 gene risk model developed for Total Therapy 2 (TT2) in the cooperative group setting.

OUTLINE:

INDUCTION THERAPY: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive dexamethasone orally (PO) once daily (QD) on days 1, 8, 15, and 22 and lenalidomide PO QD on days 1-21. Treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive dexamethasone PO QD on days 1, 2, 4, 5, 8, 9, 11, and 12; lenalidomide PO QD on days 1-14; and bortezomib intravenously (IV) over 3-5 seconds on days 1, 4, 8, and 11. Treatment repeats every 21 days for 8 courses in the absence of disease progression or unacceptable toxicity.

In both arms, patients who intend to undergo transplantation at relapse undergo peripheral blood stem cell collection, preferably after course 2.

MAINTENANCE THERAPY: After the completion of at least 4 courses (Arm I) or at least 6 courses (Arm II) of induction therapy, patients receive maintenance therapy comprising dexamethasone PO QD on days 1, 8, 15, and 22 and lenalidomide PO QD on days 1-21. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up periodically for up to 6 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have newly diagnosed multiple myeloma with measurable disease; patients with non-secretory multiple myeloma (MM) based upon standard M-component criteria (i.e., measurable serum/urine M-component) are not eligible for this study; exception: patients with non-secretory MM will be eligible only if the baseline serum Freelite is elevated (Note that serum Freelite must be drawn; serum light chains are not acceptable); all tests for establishing baseline disease status must be completed within 28 days prior to registration and documented on the baseline and follow-up tumor assessment form for multiple myeloma
* Patients must have received no prior chemotherapy for this disease; patients must have received no prior radiotherapy to a large area of the pelvis (more than half of the pelvis); prior steroid treatment is allowed provided treatment was not more than 2 weeks in duration; patients must not have received any prior treatment with bortezomib or lenalidomide
* Patients must have a Zubrod performance status (PS) of 0 - 3; NOTE: patients with PS 3 are eligible only if it is documented by the treating physician that the patient's multiple myeloma is the central cause of his/her disability; patients who have a PS of 3 due to other concurrent medical conditions are not eligible for this trial
* Platelet count >= 80 x 10^3/mcL; must be obtained within 28 days prior to registration; exception: patients with biopsy-proven heavy-marrow involvement, as defined by having at least 30% marrow cellularity, with > 50% of the cells being malignant plasma cells (documented marrow results required); in this case, although there are no required lower limits of normal for the blood counts, the treating physician must use his/her medical judgment as to the appropriateness of this study therapy for these patients
* Absolute neutrophil count (ANC) >= 1 x 10^3/mcL; must be obtained within 28 days prior to registration; exception: patients with biopsy-proven heavy-marrow involvement, as defined by having at least 30% marrow cellularity, with > 50% of the cells being malignant plasma cells (documented marrow results required); in this case, although there are no required lower limits of normal for the blood counts, the treating physician must use his/her medical judgment as to the appropriateness of this study therapy for these patients
* Hemoglobin (including patients who have been either transfused or treated with erythropoietin [EPO]) >= 9 g/dL; must be obtained within 28 days prior to registration; exception: patients with biopsy-proven heavy-marrow involvement, as defined by having at least 30% marrow cellularity, with > 50% of the cells being malignant plasma cells (documented marrow results required); in this case, although there are no required lower limits of normal for the blood counts, the treating physician must use his/her medical judgment as to the appropriateness of this study therapy for these patients
* Patients must be offered participation in the Myeloma Specimen Repository for banking and future research; with the patient's consent, bone marrow aspirates and serum specimens will be submitted to the Myeloma Specimen Repository for additional testing and banking (including SNP testing); patient consent must be obtained before specimens may be submitted
* Patients must have baseline skeletal survey to include lateral skull, anterior-posterior (AP) pelvis and posterior-anterior (PA) chest within 28 days prior to registration
* Institutions must submit a local cytogenetics report and fluorescence in situ hybridization (FISH) analysis report obtained prior to enrollment to S0777; for FISH analysis two probes will be utilized: LSI 13 (RBI) 13q14 SpectrumOrange Probe for detection of chromosome 13 deletion and LSI p53 (17p13.1) SpectrumOrange probe for detection of tumor protein (p)53 locus on chromosome 17; if these exact probes are not available locally, it is acceptable to submit results using local protocol; this must be noted on the prestudy form; NOTE: it is not required that the results of the FISH analysis be known prior to registration, only that pre-registration specimens be drawn and sent for analysis prior to registration, and the FISH analysis report be submitted
* Patients with pathologic fractures, pneumonia at diagnosis or symptomatic hyperviscosity must have these conditions attended to prior to registration (i.e., intramedullary rod, I.V. antibiotics, plasmapheresis)
* Patients must have a calculated or measured creatinine clearance > 30 cc/min; measured creatinine clearance or serum creatinine used in calculation must be obtained within 28 days prior to registration
* Patients must not have uncontrolled, active infection requiring intravenous antibiotics, New York Heart Association (NYHA) class III or class IV heart failure, myocardial infarction within the last 6 months, history of treatment for clinically significant ventricular cardiac arrhythmias, poorly controlled hypertension, or poorly controlled diabetes mellitus; patients must have undergone an electrocardiogram (EKG) within 28 days prior to registration
* Patients must not have any psychiatric illness that could potentially interfere with the completion of treatment according to this protocol
* Patients must not be hepatitis B, hepatitis C or human immunodeficiency virus (HIV) positive; patients must have a negative hepatitis B and HIV test performed within 28 days prior to registration; exception: treatment-sensitive HIV infection patients will be eligible provided that immunological and virologic indices are indicative of favorable long-term survival prospects on the basis of HIV infection, but whose life expectancy is limited predominantly by multiple myeloma rather than HIV infection in the judgment of the treating physician
* Patients must not have a history of cerebral vascular accident with persistent neurologic deficits
* Patients must be able to take aspirin 325 mg daily (or enoxaparin 40 mg subcutaneously [SQ] daily if patient is unable to take aspirin) as prophylactic anticoagulation; exception: patients receiving anticoagulation therapy such as Coumadin or heparin will NOT receive aspirin, and therefore need not be able to take it
* Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test with a sensitivity of at least 25 mIU/mL within 10 - 14 days and again within 24 hours prior to starting cycle 1 of lenalidomide; further, they must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control: one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before starting lenalidomide; FCBP must also agree to ongoing pregnancy testing; men must agree to use a latex condom during sexual contact with a FCBP, even if they have had a successful vasectomy; a FCBP is a sexually mature woman who: has not undergone a hysterectomy or bilateral oophorectomy; or has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months); all patients must be counseled by a trained counselor every 28 days about pregnancy precautions and risks of fetal exposure
* No prior malignancy is allowed except for adequately treated basal cell (or squamous cell) skin cancer, in situ cervical cancer or other cancer for which the patient has been disease-free for five years
* Patients must be offered participation in gene expression profiling (GEP) molecular studies for the evaluation of genetic polymorphisms
* All patients must be informed of the investigational nature of this study and must sign and give written consent in accordance with institutional federal guidelines
* At the time of patient registration, the treating institution's name and identification (ID) number must be provided to the statistical center in order to ensure that the current (within 365 days) date of institutional review board approval for this study has been entered into the data base

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 525 (Actual)
Dates: Start 2008-07-28 (Actual); Primary Completion 2015-11-05 (Actual); Study Completion 2026-09-18 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Brian M Durie, Principal Investigator — SWOG Cancer Research Network
Locations (499):
- United States (497):
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - University of Arizona Cancer Center-Orange Grove Campus, Tucson, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Kaiser Permanente-Deer Valley Medical Center, Antioch, California
  - PCR Oncology, Arroyo Grande, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Mills-Peninsula Medical Center, Burlingame, California
  - Kaiser Permanente-Fremont, Fremont, California
  - Kaiser Permanente-Fresno, Fresno, California
  - Saint Jude Medical Center, Fullerton, California
  - Marin General Hospital, Greenbrae, California
  - Fremont - Rideout Cancer Center, Marysville, California
  - Providence Holy Cross Medical Center, Mission Hills, California
  - Palo Alto Medical Foundation-Camino Division, Mountain View, California
  - Sutter Cancer Research Consortium, Novato, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Saint Joseph Hospital - Orange, Orange, California
  - Desert Regional Medical Center, Palm Springs, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Valley Medical Oncology Consultants, Pleasanton, California
  - Eisenhower Medical Center, Rancho Mirage, California
  - Kaiser Permanente-Redwood City, Redwood City, California
  - Kaiser Permanente-Richmond, Richmond, California
  - Kaiser Permanente-Roseville, Roseville, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - Kaiser Permanente Sacramento Medical Center, Sacramento, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Kaiser Permanente-San Rafael, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Kaiser Permanente-Stockton, Stockton, California
  - Gene Upshaw Memorial Tahoe Forest Cancer Center, Truckee, California
  - Kaiser Permanente Medical Center-Vacaville, Vacaville, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - The Medical Center of Aurora, Aurora, Colorado
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - Boulder Community Foothills Hospital, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Denver Health Medical Center, Denver, Colorado
  - Kaiser Permanente-Franklin, Denver, Colorado
  - AdventHealth Porter, Denver, Colorado
  - University of Colorado, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Saint Joseph Hospital - Cancer Centers of Colorado, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Western States Cancer Research NCORP, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Saint Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - Banner North Colorado Medical Center, Greeley, Colorado
  - Kaiser Permanente-Rock Creek, Lafayette, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Banner North Colorado Medical Center - Loveland Campus, Loveland, Colorado
  - AdventHealth Parker, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - Intermountain Health Lutheran Hospital, Wheat Ridge, Colorado
  - Danbury Hospital, Danbury, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Norwalk Hospital, Norwalk, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Mayo Clinic in Florida, Jacksonville, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - Martin Medical Center, Stuart, Florida
  - Robert and Carol Weissman Cancer Center at Martin Health, Stuart, Florida
  - Martin Hospital South, Stuart, Florida
  - Piedmont Hospital, Atlanta, Georgia
  - Atlanta Regional CCOP, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - WellStar Cobb Hospital, Austell, Georgia
  - John B Amos Cancer Center, Columbus, Georgia
  - Emory Decatur Hospital, Decatur, Georgia
  - Piedmont Fayette Hospital, Fayetteville, Georgia
  - Northside Hospital - Gwinnett, Lawrenceville, Georgia
  - Wellstar Kennestone Hospital, Marietta, Georgia
  - Southern Regional Medical Center, Riverdale, Georgia
  - Harbin Clinic Medical Oncology and Clinical Research, Rome, Georgia
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kaiser Permanente Moanalua Medical Center, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Castle Medical Center, Kailua, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Maui Memorial Medical Center, Wailuku, Hawaii
  - Pacific Cancer Institute of Maui, Wailuku, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - OSF Saint Anthony's Health Center, Alton, Illinois
  - Rush-Copley Medical Center, Aurora, Illinois
  - MacNeal Hospital and Cancer Center, Berwyn, Illinois
  - OSF Saint Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Graham Hospital Association, Canton, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Hematology and Oncology Associates, Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Heartland Cancer Research NCORP, Decatur, Illinois
  - Advocate Good Samaritan Hospital, Downers Grove, Illinois
  - Eureka Hospital, Eureka, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Illinois CancerCare-Havana, Havana, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hematology Oncology Associates of Illinois-Highland Park, Highland Park, Illinois
  - Hopedale Medical Complex - Hospital, Hopedale, Illinois
  - Midwest Center for Hematology Oncology, Joliet, Illinois
  - Duly Health and Care Joliet, Joliet, Illinois
  - Presence Saint Mary's Hospital, Kankakee, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - AMG Libertyville - Oncology, Libertyville, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Mcdonough District Hospital, Macomb, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Holy Family Medical Center, Monmouth, Illinois
  - Illinois CancerCare-Monmouth, Monmouth, Illinois
  - SSM Health Good Samaritan, Mount Vernon, Illinois
  - DuPage Medical Group-Ogden, Naperville, Illinois
  - Illinois Cancer Specialists-Niles, Niles, Illinois
  - Carle BroMenn Medical Center, Normal, Illinois
  - Carle Cancer Institute Normal, Normal, Illinois
  - Illinois CancerCare-Community Cancer Center, Normal, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Ottawa Regional Hospital and Healthcare Center, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin, Pekin, Illinois
  - Pekin Hospital, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois Valley Hospital, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - Hematology Oncology Associates of Illinois - Skokie, Skokie, Illinois
  - Illinois CancerCare-Spring Valley, Spring Valley, Illinois
  - Saint Margaret's Hospital, Spring Valley, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Northwestern Medicine Central DuPage Hospital, Winfield, Illinois
  - Franciscan Saint Francis Health-Beech Grove, Beech Grove, Indiana
  - Elkhart Clinic, Elkhart, Indiana
  - Michiana Hematology Oncology PC-Elkhart, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Fort Wayne Medical Oncology and Hematology Inc-Parkview, Fort Wayne, Indiana
  - Goshen Center for Cancer Care, Goshen, Indiana
  - Community Howard Regional Health, Kokomo, Indiana
  - IU Health La Porte Hospital, La Porte, Indiana
  - Franciscan Saint Anthony Health-Michigan City, Michigan City, Indiana
  - Michiana Hematology Oncology PC-Mishawaka, Mishawaka, Indiana
  - Saint Joseph Regional Medical Center-Mishawaka, Mishawaka, Indiana
  - The Community Hospital, Munster, Indiana
  - Michiana Hematology Oncology PC-Plymouth, Plymouth, Indiana
  - Reid Health, Richmond, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - Michiana Hematology Oncology PC-Westville, Westville, Indiana
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Iowa-Wide Oncology Research Coalition NCORP, Des Moines, Iowa
  - Mercy Medical Center - North Iowa, Mason City, Iowa
  - Ottumwa Regional Health Center, Ottumwa, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Mercy Medical Center-Sioux City, Sioux City, Iowa
  - Saint Luke's Regional Medical Center, Sioux City, Iowa
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Saint Luke's South Hospital, Overland Park, Kansas
  - Kansas City NCI Community Oncology Research Program, Prairie Village, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - AdventHealth Shawnee Mission, Shawnee Mission, Kansas
  - Cotton O'Neil Cancer Center / Stormont Vail Health, Topeka, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Wichita NCI Community Oncology Research Program, Wichita, Kansas
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Louisiana State University Health Science Center, New Orleans, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - Eastern Maine Medical Center, Bangor, Maine
  - York Hospital, York Village, Maine
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Christiana Care - Union Hospital, Elkton, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Commonwealth Hematology Oncology PC-Concord, Concord, Massachusetts
  - Dana Farber Community Cancer Care-Haverhill, Haverhill, Massachusetts
  - Dana Farber-Merrimack Valley, Methuen, Massachusetts
  - Dana Farber Community Cancer Care-Quincy, Quincy, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - Dana Farber Community Cancer Care-Stoneham, Stoneham, Massachusetts
  - Dana Farber Community Cancer Care-Weymouth, Weymouth, Massachusetts
  - Commonwealth Hematology Oncology PC-Worcester, Worcester, Massachusetts
  - Bixby Medical Center, Adrian, Michigan
  - Hickman Cancer Center, Adrian, Michigan
  - Michigan Cancer Research Consortium NCORP, Ann Arbor, Michigan
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Spectrum Health Big Rapids Hospital, Big Rapids, Michigan
  - Corewell Health Dearborn Hospital, Dearborn, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - OSF Saint Francis Hospital and Medical Group, Escanaba, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Regional Medical Center-West Flint Campus, Flint, Michigan
  - Cancer Research Consortium of West Michigan NCORP, Grand Rapids, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - Holland Community Hospital, Holland, Michigan
  - Allegiance Health, Jackson, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Beacon Kalamazoo, Kalamazoo, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - UP Health System Marquette, Marquette, Michigan
  - Mercy Memorial Hospital, Monroe, Michigan
  - Toledo Clinic Cancer Centers-Monroe, Monroe, Michigan
  - McLaren Cancer Institute-Macomb, Mount Clemens, Michigan
  - Mercy Health Partners-Hackley Campus, Muskegon, Michigan
  - Trinity Health Muskegon Hospital, Muskegon, Michigan
  - Corewell Health Lakeland Hospitals - Niles Hospital, Niles, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - Corewell Health William Beaumont University Hospital, Royal Oak, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - Corewell Health Lakeland Hospitals - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Corewell Health Lakeland Hospitals - Saint Joseph Hospital, Saint Joseph, Michigan
  - Henry Ford Health Providence Southfield Hospital, Southfield, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Henry Ford Health Warren Hospital, Warren, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Medini, Eitan MD (UIA Investigator), Alexandria, Minnesota
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Etzell, Paul S MD (UIA Investigator), Fergus Falls, Minnesota
  - Swenson, Wade II, MD (UIA Investigator), Fergus Falls, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Meeker County Memorial Hospital, Litchfield, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Virginia Piper Cancer Institute, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Saint Cloud Hospital, Saint Cloud, Minnesota
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - Saint Joseph's Hospital - Healtheast, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Woodwinds Health Campus, Woodbury, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Keesler Medical Center, Keesler Air Force Base, Mississippi
  - Singing River Hospital, Pascagoula, Mississippi
  - Southeast Missouri Hospital, Cape Girardeau, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Freeman Health System, Joplin, Missouri
  - University Health Truman Medical Center, Kansas City, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Saint Joseph Health Center, Kansas City, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - Heartland Hematology and Oncology Associates Incorporated, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Liberty Hospital, Liberty, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Mercy Infusion Center - Chippewa, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Saint Louis-Cape Girardeau CCOP, St Louis, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Montana Cancer Consortium NCORP, Billings, Montana
  - Saint Vincent Frontier Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Berdeaux, Donald MD (UIA Investigator), Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Glacier Oncology PLLC, Kalispell, Montana
  - Kalispell Medical Oncology, Kalispell, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Montana Cancer Specialists, Missoula, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Center, Missoula, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Nevada Cancer Research Foundation NCORP, Las Vegas, Nevada
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - CentraState Medical Center, Freehold, New Jersey
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Rutgers New Jersey Medical School, Newark, New Jersey
  - Lovelace Medical Center-Saint Joseph Square, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Memorial Medical Center-Las Cruces, Las Cruces, New Mexico
  - San Juan Regional Medical Center, San Juan, New Mexico
  - Adirondack Cancer Center, Glens Falls, New York
  - Garnet Health Medical Center, Middletown, New York
  - NYU Langone Hospital - Long Island, Mineola, New York
  - Mount Sinai Union Square, New York, New York
  - Mount Sinai West, New York, New York
  - Highland Hospital, Rochester, New York
  - University of Rochester, Rochester, New York
  - Montefiore Medical Center-Wakefield Campus, The Bronx, New York
  - Mission Hospital, Asheville, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - ECU Health Oncology Kinston, Kinston, North Carolina
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Southeast Clinical Oncology Research Consortium NCORP, Winston-Salem, North Carolina
  - Mid Dakota Clinic, Bismarck, North Dakota
  - Saint Alexius Medical Center, Bismarck, North Dakota
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Cleveland Clinic Cancer Center Beachwood, Beachwood, Ohio
  - Toledo Clinic Cancer Centers-Bowling Green, Bowling Green, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - North Coast Cancer Care-Clyde, Clyde, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Dayton Veterans Affairs Medical Center, Dayton, Ohio
  - Dayton NCI Community Oncology Research Program, Dayton, Ohio
  - Hematology Oncology Center Incorporated, Elyria, Ohio
  - Mercy Cancer Center-Elyria, Elyria, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Cleveland Clinic Cancer Center Independence, Independence, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Saint Rita's Medical Center, Lima, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Saint Luke's Hospital, Maumee, Ohio
  - Toledo Clinic Cancer Centers-Maumee, Maumee, Ohio
  - Toledo Radiation Oncology at Northwest Ohio Onocolgy Center, Maumee, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - Fisher-Titus Medical Center, Norwalk, Ohio
  - Saint Charles Hospital, Oregon, Ohio
  - Toledo Clinic Cancer Centers-Oregon, Oregon, Ohio
  - University Hospitals Parma Medical Center, Parma, Ohio
  - North Coast Cancer Care, Sandusky, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - Mercy Health - Saint Vincent Hospital, Toledo, Ohio
  - University of Toledo, Toledo, Ohio
  - Toledo Community Hospital Oncology Program CCOP, Toledo, Ohio
  - Mercy Health - Saint Anne Hospital, Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Clinton Memorial Hospital/Foster J Boyd Regional Cancer Center, Wilmington, Ohio
  - Cleveland Clinic Wooster Family Health and Surgery Center, Wooster, Ohio
  - Greene Memorial Hospital, Xenia, Ohio
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Adventist Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Compass Oncology Rose Quarter, Portland, Oregon
  - Legacy Emanuel Hospital and Health Center, Portland, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Butler Memorial Hospital, Butler, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Oncology Hematology Associates of Northern Pennsylvania, DuBois, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Mount Nittany Medical Center, State College, Pennsylvania
  - Associates In Hematology Oncology PC-Upland, Upland, Pennsylvania
  - Jennersville Regional Hospital, West Grove, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Geisinger South Wilkes-Barre, Wilkes-Barre, Pennsylvania
  - Hematology and Oncology Associates of Rhode Island Inc, Cranston, Rhode Island
  - Memorial Hospital of Rhode Island, Pawtucket, Rhode Island
  - Kent Hospital, Warwick, Rhode Island
  - AnMed Health Hospital, Anderson, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Medical X-Ray Center, Sioux Falls, South Dakota
  - Avera McKennan Hospital and University Health Center, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Erlanger Medical Center, Chattanooga, Tennessee
  - Jackson-Madison County General Hospital, Jackson, Tennessee
  - The Jackson Clinic PA, Jackson, Tennessee
  - Wellmont Holston Valley Hospital and Medical Center, Kingsport, Tennessee
  - University of Tennessee Health Science Center, Memphis, Tennessee
  - The Don and Sybil Harrington Cancer Center, Amarillo, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Baylor Saint Luke's Medical Center, Houston, Texas
  - Ben Taub General Hospital, Houston, Texas
  - Houston Methodist Hospital, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Michael E DeBakey VA Medical Center, Houston, Texas
  - Wilford Hall Medical Center, Lackland Air Force Base, Texas
  - Danville Regional Medical Center, Danville, Virginia
  - Fredericksburg Oncology Inc, Fredericksburg, Virginia
  - Sovah Health Martinsville, Martinsville, Virginia
  - Ballad Health Cancer Care - Norton, Norton, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Compass Oncology Vancouver, Vancouver, Washington
  - Legacy Salmon Creek Hospital, Vancouver, Washington
  - Wheeling Hospital/Schiffler Cancer Center, Wheeling, West Virginia
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Marshfield Clinic-Chippewa Center, Chippewa Falls, Wisconsin
  - HSHS Sacred Heart Hospital, Eau Claire, Wisconsin
  - Marshfield Clinic Cancer Center at Sacred Heart, Eau Claire, Wisconsin
  - Green Bay Oncology at Saint Vincent Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - University of Wisconsin Carbone Cancer Center - Johnson Creek, Johnson Creek, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Mayo Clinic Health System-Franciscan Healthcare, La Crosse, Wisconsin
  - Marshfield Medical Center - Ladysmith, Ladysmith, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Bay Area Medical Center, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Marshfield Medical Center, Marshfield, Wisconsin
  - Ascension Southeast Wisconsin Hospital - Saint Joseph Campus, Milwaukee, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - Aspirus Cancer Care - James Beck Cancer Center, Rhinelander, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - HSHS Saint Nicholas Hospital, Sheboygan, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Aspirus Cancer Care - Stevens Point, Stevens Point, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Rocky Mountain Oncology, Casper, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming
- San Juan City Hospital, San Juan, Puerto Rico
- King Faisal Specialist Hospital and Research Centre, Riyadh, Saudi Arabia

REFERENCES:
- [Derived] Banerjee R, Sexton R, Cowan AJ, Rosenberg AS, Ailawadhi S, Rajkumar SV, Kumar S, Dispenzieri A, Lonial S, Durie BGM, Richardson PG, Usmani SZ, Hoering A, Orlowski RZ. Dexamethasone dose intensity does not impact outcomes in newly diagnosed multiple myeloma: a secondary SWOG analysis. Blood. 2025 Jan 2;145(1):75-84. doi: 10.1182/blood.2024025939. PMID 39321347
- [Derived] Unger JM, LeBlanc M, Blanke CD. The Effect of Positive SWOG Treatment Trials on Survival of Patients With Cancer in the US Population. JAMA Oncol. 2017 Oct 1;3(10):1345-1351. doi: 10.1001/jamaoncol.2017.0762. PMID 28586789
- [Derived] Durie BGM, Hoering A, Abidi MH, Rajkumar SV, Epstein J, Kahanic SP, Thakuri M, Reu F, Reynolds CM, Sexton R, Orlowski RZ, Barlogie B, Dispenzieri A. Bortezomib with lenalidomide and dexamethasone versus lenalidomide and dexamethasone alone in patients with newly diagnosed myeloma without intent for immediate autologous stem-cell transplant (SWOG S0777): a randomised, open-label, phase 3 trial. Lancet. 2017 Feb 4;389(10068):519-527. doi: 10.1016/S0140-6736(16)31594-X. Epub 2016 Dec 23. PMID 28017406
- [Derived] Usmani SZ, Heuck C, Mitchell A, Szymonifka J, Nair B, Hoering A, Alsayed Y, Waheed S, Haider S, Restrepo A, Van Rhee F, Crowley J, Barlogie B. Extramedullary disease portends poor prognosis in multiple myeloma and is over-represented in high-risk disease even in the era of novel agents. Haematologica. 2012 Nov;97(11):1761-7. doi: 10.3324/haematol.2012.065698. Epub 2012 Jun 11. PMID 22689675
- See also: Data Available: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive. — https://nctn-data-archive.nci.nih.gov/

RESULTS

PARTICIPANT FLOW:
Period: Randomization & Eligibility
Arm/Group | Arm I (Dexamethasone and Lenalidomide) | Arm II (Dexamethasone, Lenalidomide, Bortezomib)
Started | 261 | 264
Eligible and Analyzable (All patients who were consented and did not withdraw consent prior to treatment are "Analyzable".) | 229 | 242
Completed ("Completed" does not apply to this study period.) | 229 | 242
Not Completed | 32 | 22
Not completed — Ineligible | 31 | 21
Not completed — Withdrew Consent prior to therapy start | 1 | 0
Not completed — Invalid Consent | 0 | 1
Period: Induction Therapy
Arm/Group | Arm I (Dexamethasone and Lenalidomide) | Arm II (Dexamethasone, Lenalidomide, Bortezomib)
Started | 229 | 242
Completed | 146 | 137
Not Completed | 83 | 105
Not completed — Adverse Event | 22 | 55
Not completed — Withdrawal by Subject | 10 | 3
Not completed — Progression/Relapse | 24 | 12
Not completed — Death | 3 | 7
Not completed — Not Protocol-Specified | 24 | 28
Period: Maintenance
Arm/Group | Arm I (Dexamethasone and Lenalidomide) | Arm II (Dexamethasone, Lenalidomide, Bortezomib)
Started | 143 (3 patients who completed induction did not continue on to maintenance due to refusal (1), other (2).) | 135 (2 patients who completed induction did not continue on to maintenance due to other (2).)
Completed (Patients were treated until progression or removal/refusal. "Completed" does not apply.) | 0 | 0
Not Completed | 143 | 135
Not completed — Adverse Event | 27 | 31
Not completed — Withdrawal by Subject | 6 | 4
Not completed — Progression/Relapse | 67 | 42
Not completed — Death | 3 | 3
Not completed — Not Protocol-Specified | 14 | 15
Not completed — On Treatment | 26 | 40

BASELINE CHARACTERISTICS:
Population: Includes all eligible and analyzable patients.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Dexamethasone and Lenalidomide) | Arm II (Dexamethasone, Lenalidomide, Bortezomib) | Total
Number analyzed (Participants) | 229 | 242 | 471
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 120 | 149 | 269
  >=65 years | 109 | 93 | 202
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 107 | 89 | 196
  Male | 122 | 153 | 275
ISS Stage [Count of Participants; unit: Participants] — International Staging System (ISS) Criteria:
  Stage I: Serum β2-microglobulin < 3.5mg/L and Serum Albumin ≥ 3.5 g/dL; expected median survival is 62 months. Stage II*: Not Stage I or III; expected median survival is 44 months. Stage III: Serum β2-microglobulin > 5.5 mg/L; expected median survival is 29 months.
  *There are two categories for stage II: serum β2-microglobulin < 3.5 mg/L but serum albumin < 3.5 g/dL; or serum β2-microglobulin 3.5 to < 5.5 mg/L irrespective of the serum albumin level.
  Participants
    ISS Stage I or II | 150 | 164 | 314
    ISS Stage III | 79 | 78 | 157

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: Unstratified median progression-free survival in months.
Time Frame: From date of registration to date of first documentation of progression or symptomatic deterioration, or death due to any cause, assessed up to 6 years
Population: All eligible and analyzable patients are included. An analyzable patient is one who provided valid consent and who did not withdraw consent prior to initiating treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm I (Dexamethasone and Lenalidomide) | Arm II (Dexamethasone, Lenalidomide, Bortezomib)
Number analyzed (Participants) | 229 | 242
Months | 30 [29 to 39] | 43 [39 to 52]
Statistical Analysis 1: Comparison: Arm I (Dexamethasone and Lenalidomide) vs Arm II (Dexamethasone, Lenalidomide, Bortezomib); With four years of patient accrual and two and a half years of follow-up, 220 patients per arm yields 87% power to detect an increase of PFS of 50%, from a median of 3 years to 4.5 years, which corresponds to a hazard ratio of 1.5. These calculations are based on a one-sided stratified log-rank test at level 0.025 with two interim analyses. The final analysis will be carried out at the 0.02 significance level to allow for two interim analyses at the 0.0025 significance level; Test type: Superiority; p = 0.0018, Log Rank — The p-value is from a one-sided, stratified log-rank test. Stratification factors include those factors by which patients were randomized: intent to transplant (yes vs no) and ISS Stage (I vs II vs III); Hazard Ratio (HR) = 0.712, 96% CI 2-sided [0.560 to 0.906] — The hazard ratio compares Bortezomib/Lenalidomide/Dexamethasone against Lenalidomide/Dexamethasone

2. Secondary Outcome: Overall Survival
Description: Unstratified median overall survival in months.
Time Frame: Up to 6 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm I (Dexamethasone and Lenalidomide) | Arm II (Dexamethasone, Lenalidomide, Bortezomib)
Number analyzed (Participants) | 229 | 242
Months | 64 [56 to NA] — The upper bound of the confidence interval has not yet been reached. | 75 [65 to NA] — The upper bound of the confidence interval has not yet been reached.
Statistical Analysis 1: Comparison: Arm I (Dexamethasone and Lenalidomide) vs Arm II (Dexamethasone, Lenalidomide, Bortezomib); Overall survival will be compared between the two treatment arms using a stratified log-rank test; Test type: Superiority; p = 0.0250, Log Rank — The p-value is based on a two-sided, stratified log rank test. Stratification factors include those factors by which patients were randomized: intent to transplant (yes vs no) and ISS Stage (I vs II vs III); Hazard Ratio (HR) = 0.709, 95% CI 2-sided [0.524 to 0.959] — The hazard ratio compares Bortezomib/Lenalidomide/Dexamethasone against Lenalidomide/Dexamethasone

3. Secondary Outcome: Response Rates ()
Description: The response rate was calculated as the number of patients with documented confirmed partial response (PR) or better, which includes confirmed/unconfirmed stringent complete response (sCR), confirmed/unconfirmed complete response (CR), confirmed/unconfirmed very good partial response (VGPR), or confirmed partial response (PR), as best response divided by the total number of evaluable patients, in each arm. Patients with measurable disease, as defined in the protocol, are evaluable. Response rates were compared between the two treatment arms using a stratified Cochran-Mantel-Haenszel test. Response designations were based on the International Uniform Response Criteria for Multiple Myeloma. Due to the complexity of these criteria, the details of these criteria have been omitted.
Time Frame: Up to 6 years
Population: All eligible, analyzable patients are included.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Dexamethasone and Lenalidomide) | Arm II (Dexamethasone, Lenalidomide, Bortezomib)
Number analyzed (Participants) | 229 | 242
Participants | 153 | 176
Statistical Analysis 1: Comparison: Arm I (Dexamethasone and Lenalidomide) vs Arm II (Dexamethasone, Lenalidomide, Bortezomib); Test type: Superiority or Other; p = 0.20, Cochran-Mantel-Haenszel — The p-value is based on a stratified Cochran-Mantel-Haenszel test. Stratification factors include those factors by which patients were randomized: intent to transplant (yes vs no) and ISS Stage (I vs II vs III)

ADVERSE EVENTS:
Description: The number at risk excludes patients who went off study prior to starting treatment and were thus not evaluated for toxicity. The adverse events reported here are current up through the time of upload of these data.
Arm/Group | Arm I (Dexamethasone and Lenalidomide) | Arm II (Dexamethasone, Lenalidomide, Bortezomib)
Serious Adverse Events (participants affected / at risk) | 105/222 | 124/237
Other Adverse Events (participants affected / at risk) | 209/222 | 232/237
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Dexamethasone and Lenalidomide) (N=222) | Arm II (Dexamethasone, Lenalidomide, Bortezomib) (N=237)
Febrile neutropenia (Blood and lymphatic system disorders) | 5 | 0
Hemoglobin (Blood and lymphatic system disorders) | 24 | 13
Hemolysis (Blood and lymphatic system disorders) | 1 | 0
Cardiac Arrhythmia-Other (Cardiac disorders) | 0 | 1
Cardiac General-Other (Cardiac disorders) | 1 | 3
Cardiac-ischemia/infarction (Cardiac disorders) | 4 | 1
Conduction abnormality NOS (Cardiac disorders) | 1 | 1
Left ventricular diastolic dysfunction (Cardiac disorders) | 4 | 1
Left ventricular systolic dysfunction (Cardiac disorders) | 4 | 0
Pain - Cardiac/heart (Cardiac disorders) | 2 | 0
SVT and nodal arrhythmia - Atrial fibrillation (Cardiac disorders) | 5 | 5
SVT and nodal arrhythmia - Atrial flutter (Cardiac disorders) | 1 | 0
SVT and nodal arrhythmia - Sinus bradycardia (Cardiac disorders) | 1 | 2
SVT and nodal arrhythmia - Sinus tachycardia (Cardiac disorders) | 1 | 0
Valvular heart disease (Cardiac disorders) | 1 | 0
Thyroid function, high (Endocrine disorders) | 0 | 1
Cataract (Eye disorders) | 1 | 0
Dry eye syndrome (Eye disorders) | 0 | 1
Ocular/Visual-Other (Eye disorders) | 0 | 1
Ophthalmoplegia/diplopia (double vision) (Eye disorders) | 0 | 1
Vision-blurred vision (Eye disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 2
Constipation (Gastrointestinal disorders) | 0 | 2
Diarrhea (Gastrointestinal disorders) | 6 | 10
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 1 | 1
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 1 | 1
Gastritis (including bile reflux gastritis) (Gastrointestinal disorders) | 1 | 0
Gastrointestinal-Other (Gastrointestinal disorders) | 0 | 2
Hemorrhage, GI - Lower GI NOS (Gastrointestinal disorders) | 1 | 4
Hemorrhage, GI - Rectum (Gastrointestinal disorders) | 2 | 1
Hemorrhage, GI - Stomach (Gastrointestinal disorders) | 0 | 1
Hemorrhage, GI - Upper GI NOS (Gastrointestinal disorders) | 0 | 1
Hemorrhage, GI - Varices (rectal) (Gastrointestinal disorders) | 1 | 0
Ileus, GI (functional obstruction of bowel) (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 2
Obstruction, GI - Colon (Gastrointestinal disorders) | 1 | 0
Obstruction, GI - Small bowel NOS (Gastrointestinal disorders) | 0 | 3
Obstruction, GI - Stomach (Gastrointestinal disorders) | 0 | 1
Pain - Abdomen NOS (Gastrointestinal disorders) | 2 | 5
Perforation, GI - Colon (Gastrointestinal disorders) | 1 | 1
Typhlitis (cecal inflammation) (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 3
Death - Multi-organ failure (General disorders) | 0 | 1
Death not associated with CTCAE term - Death NOS (General disorders) | 1 | 4
Edema: limb (General disorders) | 1 | 2
Extremity-lower (gait/walking) (General disorders) | 1 | 1
Fatigue (asthenia, lethargy, malaise) (General disorders) | 5 | 8
Fever in absence of neutropenia, ANC lt1.0x10e9/L (General disorders) | 1 | 0
Flu-like syndrome (General disorders) | 0 | 2
Pain - Chest/thorax NOS (General disorders) | 0 | 3
Pain - Pain NOS (General disorders) | 1 | 3
Pain-Other (General disorders) | 0 | 1
Sudden death (General disorders) | 1 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 2
Hepatobiliary/Pancreas-Other (Hepatobiliary disorders) | 1 | 0
Liver dysfunction/failure (clinical) (Hepatobiliary disorders) | 2 | 2
Pain - Gallbladder (Hepatobiliary disorders) | 1 | 0
Allergic reaction/hypersensitivity (Immune system disorders) | 1 | 1
Colitis, infectious (e.g., Clostridium difficile) (Infections and infestations) | 1 | 2
Inf (clin/microbio) w/Gr 3-4 neuts - Blood (Infections and infestations) | 1 | 0
Inf (clin/microbio) w/Gr 3-4 neuts - Bronchus (Infections and infestations) | 1 | 0
Inf (clin/microbio) w/Gr 3-4 neuts - Cecum (Infections and infestations) | 1 | 0
Inf (clin/microbio) w/Gr 3-4 neuts - Lung (Infections and infestations) | 3 | 3
Inf (clin/microbio) w/Gr 3-4 neuts - UTI (Infections and infestations) | 1 | 0
Inf (clin/microbio) w/Gr 3-4 neuts - Upper airway (Infections and infestations) | 1 | 0
Inf w/normal ANC or Gr 1-2 neutrophils - Bladder (Infections and infestations) | 1 | 0
Inf w/normal ANC or Gr 1-2 neutrophils - Blood (Infections and infestations) | 0 | 2
Inf w/normal ANC or Gr 1-2 neutrophils - Catheter (Infections and infestations) | 0 | 1
Inf w/normal ANC or Gr 1-2 neutrophils - Colon (Infections and infestations) | 1 | 0
Inf w/normal ANC or Gr 1-2 neutrophils - Lung (Infections and infestations) | 6 | 8
Inf w/normal ANC or Gr 1-2 neutrophils - UTI (Infections and infestations) | 1 | 5
Inf w/normal ANC or Gr 1-2 neutrophils - Wound (Infections and infestations) | 2 | 0
Infection with unknown ANC - Anal/perianal (Infections and infestations) | 0 | 1
Infection with unknown ANC - Blood (Infections and infestations) | 3 | 4
Infection with unknown ANC - Bone (osteomyelitis) (Infections and infestations) | 1 | 0
Infection with unknown ANC - Bronchus (Infections and infestations) | 0 | 1
Infection with unknown ANC - Catheter-related (Infections and infestations) | 0 | 1
Infection with unknown ANC - Eye NOS (Infections and infestations) | 1 | 0
Infection with unknown ANC - Heart (endocarditis) (Infections and infestations) | 0 | 1
Infection with unknown ANC - Joint (Infections and infestations) | 1 | 1
Infection with unknown ANC - Lung (pneumonia) (Infections and infestations) | 15 | 10
Infection with unknown ANC - Meninges (meningitis) (Infections and infestations) | 1 | 0
Infection with unknown ANC - Mucosa (Infections and infestations) | 0 | 1
Infection with unknown ANC - Pharynx (Infections and infestations) | 1 | 0
Infection with unknown ANC - Sinus (Infections and infestations) | 1 | 0
Infection with unknown ANC - Skin (cellulitis) (Infections and infestations) | 0 | 4
Infection with unknown ANC - Upper airway NOS (Infections and infestations) | 0 | 2
Infection with unknown ANC - Urinary tract NOS (Infections and infestations) | 2 | 2
Infection-Other (Infections and infestations) | 5 | 4
Fracture (Injury, poisoning and procedural complications) | 4 | 6
Thrombosis/embolism (vascular access-related) (Injury, poisoning and procedural complications) | 1 | 3
Wound complication, non-infectious (Injury, poisoning and procedural complications) | 0 | 1
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 2 | 3
AST, SGOT (Investigations) | 2 | 1
Alkaline phosphatase (Investigations) | 1 | 1
Bilirubin (hyperbilirubinemia) (Investigations) | 1 | 1
Cardiac troponin I (cTnI) (Investigations) | 0 | 1
Creatinine (Investigations) | 9 | 7
INR (of prothrombin time) (Investigations) | 1 | 3
Leukocytes (total WBC) (Investigations) | 2 | 3
Lymphopenia (Investigations) | 0 | 5
Metabolic/Laboratory-Other (Investigations) | 0 | 1
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 2 | 5
PTT (Partial thromboplastin time) (Investigations) | 0 | 1
Platelets (Investigations) | 5 | 13
Weight loss (Investigations) | 1 | 2
Acidosis (metabolic or respiratory) (Metabolism and nutrition disorders) | 0 | 1
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 2 | 5
Calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 2 | 2
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 6 | 5
Dehydration (Metabolism and nutrition disorders) | 9 | 17
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 6 | 6
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 2 | 1
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 1 | 2
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 2 | 12
Sodium, serum-high (hypernatremia) (Metabolism and nutrition disorders) | 1 | 0
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 3 | 5
Tumor lysis syndrome (Metabolism and nutrition disorders) | 2 | 2
Uric acid, serum-high (hyperuricemia) (Metabolism and nutrition disorders) | 1 | 0
Arthritis (non-septic) (Musculoskeletal and connective tissue disorders) | 1 | 2
Joint-effusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle weakness, not d/t neuropathy - Extrem-lower (Musculoskeletal and connective tissue disorders) | 1 | 4
Muscle weakness, not d/t neuropathy - body/general (Musculoskeletal and connective tissue disorders) | 3 | 11
Musculoskeletal/Soft Tissue-Other (Musculoskeletal and connective tissue disorders) | 1 | 3
Osteonecrosis (avascular necrosis) (Musculoskeletal and connective tissue disorders) | 2 | 1
Pain - Back (Musculoskeletal and connective tissue disorders) | 4 | 4
Pain - Bone (Musculoskeletal and connective tissue disorders) | 3 | 1
Pain - Chest wall (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain - Extremity-limb (Musculoskeletal and connective tissue disorders) | 1 | 2
Pain - Joint (Musculoskeletal and connective tissue disorders) | 1 | 1
Pain - Muscle (Musculoskeletal and connective tissue disorders) | 1 | 0
Death - Disease progression NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Myelodysplasia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Secondary Malignancy-poss rel to cancer Tx (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2
CNS cerebrovascular ischemia (Nervous system disorders) | 3 | 1
Cognitive disturbance (Nervous system disorders) | 2 | 0
Dizziness (Nervous system disorders) | 0 | 4
Encephalopathy (Nervous system disorders) | 3 | 1
Hemorrhage, CNS (Nervous system disorders) | 1 | 0
Neurology-Other (Nervous system disorders) | 3 | 1
Neuropathy: motor (Nervous system disorders) | 1 | 2
Neuropathy: sensory (Nervous system disorders) | 2 | 7
Ocular/Visual-Other (Nervous system disorders) | 0 | 1
Pain - Head/headache (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 0 | 2
Somnolence/depressed level of consciousness (Nervous system disorders) | 3 | 2
Syncope (fainting) (Nervous system disorders) | 5 | 12
Taste alteration (dysgeusia) (Nervous system disorders) | 1 | 0
Tremor (Nervous system disorders) | 0 | 2
Confusion (Psychiatric disorders) | 5 | 3
Mood alteration - depression (Psychiatric disorders) | 0 | 1
Psychosis (hallucinations/delusions) (Psychiatric disorders) | 1 | 0
Fistula, GU - Bladder (Renal and urinary disorders) | 0 | 1
Glomerular filtration rate (Renal and urinary disorders) | 1 | 1
Hemorrhage, GU - Urinary NOS (Renal and urinary disorders) | 1 | 0
Incontinence, urinary (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 13 | 3
Renal/Genitourinary-Other (Renal and urinary disorders) | 2 | 2
Urinary retention (including neurogenic bladder) (Renal and urinary disorders) | 1 | 1
Adult respiratory distress syndrome (ARDS) (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Bronchospasm, wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 4 | 9
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 | 6
Mucositis/stomatitis (clinical exam) - Pharynx (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pain - Pleura (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 3 | 6
Pulmonary/Upper Respiratory-Other (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Rash/desquamation (Skin and subcutaneous tissue disorders) | 2 | 1
Skin breakdown/decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (hives, welts, wheals) (Skin and subcutaneous tissue disorders) | 0 | 1
Hypertension (Vascular disorders) | 2 | 4
Hypotension (Vascular disorders) | 2 | 16
Thrombosis/thrombus/embolism (Vascular disorders) | 9 | 8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Dexamethasone and Lenalidomide) (N=222) | Arm II (Dexamethasone, Lenalidomide, Bortezomib) (N=237)
Hemoglobin (Blood and lymphatic system disorders) | 162 | 172
Tinnitus (Ear and labyrinth disorders) | 19 | 9
Cataract (Eye disorders) | 14 | 19
Dry eye syndrome (Eye disorders) | 13 | 19
Vision-blurred vision (Eye disorders) | 41 | 53
Constipation (Gastrointestinal disorders) | 119 | 141
Diarrhea (Gastrointestinal disorders) | 99 | 113
Distention/bloating, abdominal (Gastrointestinal disorders) | 8 | 13
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 27 | 30
Flatulence (Gastrointestinal disorders) | 24 | 22
Gastrointestinal-Other (Gastrointestinal disorders) | 12 | 10
Heartburn/dyspepsia (Gastrointestinal disorders) | 43 | 58
Mucositis/stomatitis (clinical exam) - Oral cavity (Gastrointestinal disorders) | 20 | 16
Mucositis/stomatitis (functional/symp) - Oral cav (Gastrointestinal disorders) | 11 | 17
Nausea (Gastrointestinal disorders) | 88 | 105
Pain - Abdomen NOS (Gastrointestinal disorders) | 33 | 43
Pain - Dental/teeth/peridontal (Gastrointestinal disorders) | 13 | 6
Vomiting (Gastrointestinal disorders) | 38 | 47
Edema: limb (General disorders) | 90 | 114
Extremity-lower (gait/walking) (General disorders) | 15 | 15
Fatigue (asthenia, lethargy, malaise) (General disorders) | 178 | 191
Fever in absence of neutropenia, ANC lt1.0x10e9/L (General disorders) | 37 | 48
Pain - Chest/thorax NOS (General disorders) | 11 | 15
Pain-Other (General disorders) | 36 | 43
Rigors/chills (General disorders) | 28 | 34
Inf w/normal ANC or Gr 1-2 neutrophils - Lung (Infections and infestations) | 21 | 20
Inf w/normal ANC or Gr 1-2 neutrophils - Skin (Infections and infestations) | 15 | 11
Inf w/normal ANC or Gr 1-2 neutrophils - Up airway (Infections and infestations) | 17 | 20
Infection-Other (Infections and infestations) | 13 | 29
Bruising (in absence of Gr 3-4 thrombocytopenia) (Injury, poisoning and procedural complications) | 23 | 24
Fracture (Injury, poisoning and procedural complications) | 8 | 15
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 59 | 70
AST, SGOT (Investigations) | 50 | 71
Alkaline phosphatase (Investigations) | 50 | 68
Bilirubin (hyperbilirubinemia) (Investigations) | 23 | 34
Creatinine (Investigations) | 78 | 69
Leukocytes (total WBC) (Investigations) | 137 | 124
Lymphopenia (Investigations) | 72 | 76
Metabolic/Laboratory-Other (Investigations) | 20 | 24
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 117 | 91
Platelets (Investigations) | 130 | 144
Weight gain (Investigations) | 22 | 17
Weight loss (Investigations) | 59 | 62
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 79 | 86
Anorexia (Metabolism and nutrition disorders) | 77 | 92
Calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 28 | 17
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 122 | 130
Dehydration (Metabolism and nutrition disorders) | 19 | 26
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 140 | 138
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 25 | 40
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 30 | 32
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 33 | 24
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 25 | 15
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 81 | 92
Sodium, serum-high (hypernatremia) (Metabolism and nutrition disorders) | 17 | 20
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 66 | 84
Muscle weakness, not d/t neuropathy - Extrem-lower (Musculoskeletal and connective tissue disorders) | 15 | 13
Muscle weakness, not d/t neuropathy - body/general (Musculoskeletal and connective tissue disorders) | 47 | 57
Musculoskeletal/Soft Tissue-Other (Musculoskeletal and connective tissue disorders) | 22 | 20
Pain - Back (Musculoskeletal and connective tissue disorders) | 91 | 97
Pain - Bone (Musculoskeletal and connective tissue disorders) | 36 | 44
Pain - Chest wall (Musculoskeletal and connective tissue disorders) | 11 | 19
Pain - Extremity-limb (Musculoskeletal and connective tissue disorders) | 51 | 73
Pain - Joint (Musculoskeletal and connective tissue disorders) | 66 | 58
Pain - Muscle (Musculoskeletal and connective tissue disorders) | 51 | 62
Pain - Neck (Musculoskeletal and connective tissue disorders) | 20 | 17
Dizziness (Nervous system disorders) | 71 | 86
Memory impairment (Nervous system disorders) | 5 | 14
Neurology-Other (Nervous system disorders) | 15 | 6
Neuropathy: motor (Nervous system disorders) | 23 | 52
Neuropathy: sensory (Nervous system disorders) | 112 | 173
Pain - Head/headache (Nervous system disorders) | 35 | 45
Pain - Neuralgia/peripheral nerve (Nervous system disorders) | 5 | 13
Taste alteration (dysgeusia) (Nervous system disorders) | 56 | 71
Tremor (Nervous system disorders) | 30 | 25
Confusion (Psychiatric disorders) | 20 | 18
Insomnia (Psychiatric disorders) | 94 | 99
Mood alteration - anxiety (Psychiatric disorders) | 43 | 37
Mood alteration - depression (Psychiatric disorders) | 45 | 41
Glomerular filtration rate (Renal and urinary disorders) | 12 | 14
Proteinuria (Renal and urinary disorders) | 15 | 13
Urinary frequency/urgency (Renal and urinary disorders) | 16 | 12
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 35 | 28
Cough (Respiratory, thoracic and mediastinal disorders) | 77 | 93
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 86 | 86
Hemorrhage, pulmonary/upper respiratory - Nose (Respiratory, thoracic and mediastinal disorders) | 19 | 16
Nasal cavity/paranasal sinus reactions (Respiratory, thoracic and mediastinal disorders) | 13 | 22
Pain - Throat/pharynx/larynx (Respiratory, thoracic and mediastinal disorders) | 6 | 13
Pulmonary/Upper Respiratory-Other (Respiratory, thoracic and mediastinal disorders) | 14 | 14
Voice changes/dysarthria (Respiratory, thoracic and mediastinal disorders) | 8 | 19
Dermatology/Skin-Other (Skin and subcutaneous tissue disorders) | 23 | 16
Dry skin (Skin and subcutaneous tissue disorders) | 45 | 41
Hair loss/Alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 14 | 20
Pruritus/itching (Skin and subcutaneous tissue disorders) | 45 | 23
Rash/desquamation (Skin and subcutaneous tissue disorders) | 57 | 56
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 9 | 17
Sweating (diaphoresis) (Skin and subcutaneous tissue disorders) | 27 | 29
Flushing (Vascular disorders) | 27 | 17
Hot flashes/flushes (Vascular disorders) | 16 | 14
Hypertension (Vascular disorders) | 37 | 35
Hypotension (Vascular disorders) | 18 | 27
Thrombosis/thrombus/embolism (Vascular disorders) | 21 | 22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less